CLINICAL TRIAL: NCT05741034
Title: Multicenter, Evaluator-blinded, Randomized, Controlled Study of the Safety and Effectiveness of JUVÉDERM® VOLITE™ for Correction of Neck Lines in Chinese Adults
Brief Title: A Study to Assess Adverse Events and Effectiveness of Injected JUVÉDERM® VOLITE™ Gel Filler for Change in Neck Lines in Adult Chinese Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M21-870
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Neck Lines
Keywords: Neck Lines; Skin Wrinkling; Juvederm VOLITE; VOLITE

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JUVÉDERM® VOLITE™ (Experimental): Participants will receive VOLITE for initial treatment and exit the study at month 12 after last treatment.
  Participants may have the opportunity to receive optional touch-up treatment of VOLITE during the follow-up duration period.
  Interventions: Device: JUVÉDERM® VOLITE™
- Control - No Treatment (Other): Participants in the control group will receive no treatment. At Month 2, these participants will have the option to receive VOLITE treatment and exit the study at month 9 after last treatment.
  Interventions: Device: JUVÉDERM® VOLITE™; Other: Control

INTERVENTIONS:
Device: JUVÉDERM® VOLITE™ — Injection, subdermal and/or intradermal
  Other Names: AGN-8015
Other: Control — No-treatment control
  Arms: Control - No Treatment

SUMMARY:
The cumulative effect of aging and environmental exposures (ie, ultraviolet, infrared, and visible light radiation and pollution) leads to wrinkles, discoloration, laxity, and roughness of sun exposed skin. The neck is a frequently mentioned area by participants complaining about its crepey texture and deep lines. JUVÉDERM® VOLITE™ is a crosslinked Hyaluronic Acid (HA) gel implant formulated with lidocaine that was developed to provide a safe, minimally invasive method of treating fine lines and improving skin quality. The purpose of this study is to assess adverse events and effectiveness of VOLITE in Chinese adults seeking correction of transverse neck lines.

VOLITE is an investigational product being developed for correction of transverse neck lines. Participants are placed in 1 of 2 groups, called treatment arms. There is a 1 in 3 chance that participants will be assigned to the control group. Around 159 adult participants with transverse neck lines will be enrolled in the study at approximately 8 sites in China.

Participants in the treatment group will receive the initial injection of VOLITE at Visit 1 and followed for up to 13 months. Participants may have the opportunity to receive optional touch-up treatment of VOLITE during the follow-up duration period. Participants in the control group will receive no treatment but will have the opportunity to receive VOLITE treatment after 2 months. Participants in the control group will be followed for up to 10 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants in general good health as determined by Treating Investigator's (TI) judgment, including no known active pandemic infection.
* Participants seeking improvement of transverse neck lines and hydration in neck area.
* Has moderate or severe transverse neck lines (ATNLS Grade 2 or 3) on EI live assessment.
* The participant is able to achieve at least a 1-point improvement in Allergan Transverse Neck Lines Scale (ATNLS) score with the allowed injection volume in the judgment of TI.

Exclusion Criteria:

* Neck deformity or significant skin laxity with severe redundant folds.
* History of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), HA (hyaluronic acid) products, or Streptococcal protein, or is planning to undergo desensitization therapy during the study.
* Have a history of or currently suffer from autoimmune disease (e.g., rheumatoid arthritis, Crohn's disease).
* Current cutaneous inflammatory or infectious processes (e.g., acne, herpes, dermatitis), abscess, an unhealed wound, or a cancerous or precancerous lesion on skin of the neck.
* History of thyroid cancer, thyroid-related diseases, skin cancer of the neck, radiation of the treatment area, or de novo cancer in the treatment area.
* Tendency to develop hypertrophic scarring.
* Has ever received permanent soft tissue fillers (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene), calcium hydroxyapatite filler, or autologous fat in the neck area.
* Has undergone neck surgery.
* Semi-permanent soft tissue fillers (e.g., poly-L-lactic acid, polycaprolactone) in the neck area within 2 years before enrollment.
* Botulinum toxin in the neck area within 6 months before enrollment.
* Neck tattoos, piercings, pigmentation, hair, or past trauma that would interfere with the visualization of the neck area for the effectiveness assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" status based on Evaluating Investigator's (EI) live assessment of transverse neck lines using the Allergan Transverse Neck Lines Scale (ATNLS) | Month 2
  A "responder" is a participant with at least 1-grade improvement on the ATNLS. ATNLS is a 5-point photonumeric scale to grade the severity of transverse neck lines (0=None, 4=Extreme).
Number of Participants with Adverse Events | Up to 13 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for EI's Assessment of global aesthetic improvement on the neck using the Global Aesthetic Improvement Scale (GAIS) | Month 2
  A "responder" is a participant who shows improvement in the overall aesthetic assessment on the neck using GAIS. GAIS is a 5-point ordinal scale (2=Much Improved, -2=Much Worse).
Percentage of Participants Achieving "Responder" Status for Participant's Assessment of global aesthetic improvement on the Neck using GAIS | Month 2
  A "responder" is a participant who shows improvement in the overall aesthetic assessment in the neck using GAIS. GAIS is a 5-point ordinal scale (2=Much Improved, -2=Much Worse)
Change from baseline to Month 2 on FACE-Q Appraisal of Neck questionnaire overall score | Baseline to Month 2
  FACE-Q is a 10-item questionnaire assessing various aspects of the neck appearance. In the FACE-Q Appraisal of Neck Lines questionnaire, the responses will be summed and converted to a Rasch-transformed score that ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (9):
- China (9):
  - China-Japan Friendship Hospital /ID# 243984, Beijing, Beijing Municipality
  - Beijing Hospital /ID# 243982, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 243980, Xicheng District, Beijing Municipality
  - The Third Affiliated Hospital, Sun Yat-Sen University /ID# 243987, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 243981, Wuhan, Hubei
  - Zhongda Hospital Southeast University /ID# 243986, Nanjing, Jiangsu
  - Wuxi People's Hospital /ID# 245875, Wuxi, Jiangsu
  - Huashan Hospital, Fudan University /ID# 244044, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital /ID# 244107, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M21-870#additional-resources-section